CLINICAL TRIAL: NCT02835352
Title: Impact of Essential Oils on Anxiety of Patients Suffering From Metastasis Cancer - Feasibility Study
Brief Title: Essential Oils on Anxiety of Patients Suffering From Cancer
Acronym: RHECAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow recruitment and study data to be recorded not available.
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-AH-DOUL-SC
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Neoplasm Metastasis
Keywords: anxiety
MeSH Terms: conditions — Neoplasm Metastasis; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Essential oils then oil massages (Experimental): Essential oils massages will be done as needed during a period of 7 days, then oïl massages as needed will be done during a follow-up period of 7 days
  Interventions: Other: Essential oils massages; Other: Oil massages
- Oil then essential oils massages (Experimental): Oil massages will be done as needed during a period of 7 days, then essential oïl massages as needed will be done during a follow-up period of 7 days
  Interventions: Other: Essential oils massages; Other: Oil massages

INTERVENTIONS:
Other: Essential oils massages
Other: Oil massages

SUMMARY:
This study evaluates the impact of essential oils massage on anxiety of patients who are suffering from cancer at a metastasis stage. Half of patients will be massaged first by essential oils and then by oil only. The other half will be massaged first by oil and then by essential oils.

ELIGIBILITY:
Inclusion Criteria:

* Adult suffering from cancer at a metastatic stage
* Life expectancy > 15 days, assessed by investigator
* Hospitalized at the Chevrel unit from Centre Eugène Marquis, palliative unit care, for more than 15 days
* Regular anxiolytic treatment or imperative need to introduce anxiolytic treatment (assessed by investigator) within 48 hours following his hospitalization entry
* > 18 years

Exclusion Criteria:

* Patient already recruited in a therapeutic trial
* Patient not covered by a social security system
* Pregnant or likely pregnant patient, breastfeeding patient
* Allergy to any component of essential oils mixture and vegetable oils : bitter orange petitgrain, fine lavender, ylang-ylang, macadamia
* Minors, people deprived of their liberty or protected people,
* Impaired cognitive functions making impossible to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Anxiolytic consumption | 7 days
  Anxiolytic consumption will be assessed at day 7 at the end of each phase

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Hutin, MD, Principal Investigator — Centre Eugène Marquis
Locations (1):
- Centre Eugène Marquis, Rennes, France

IPD SHARING:
Plan to Share IPD: No
Not authorized by French law